CLINICAL TRIAL: NCT03077659
Title: Phase IIa Dose Escalation Trial of NanoPac® Focal Therapy for Prostate Cancer in Subjects Undergoing Radical Prostatectomy
Brief Title: Trial of NanoPac® Focal Therapy in Subjects With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2016-02
Record Dates: First submitted 2017-02-28; First posted 2017-03-13 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: prostate cancer; prostatic neoplasms; genital neoplasms, male; urogenital neoplasms; prostatic diseases
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Prostatic Diseases | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Open-label, dose rising, Phase IIa trial. The study will include a dose escalation phase and a dose confirmation phase. In the dose escalation phase, NanoPac® concentrations of 6, 10, and 15 mg/mL in an injection volume of 20% of the lobe of the prostate containing the dominant lesion will be studied in cohorts of 3, with cohorts enrolled sequentially starting at the lowest concentration. Following DSMB review of the cohort data the next cohort may begin enrolling, or an additional 3 at the current dose may be enrolled, or if the first dose does not provide adequate safety and tolerability the study may be halted. The dose determined to be the most suitable for further evaluation, defined as the highest dose with an acceptable safety and tolerability profile as determined by the DSMB, will enroll additional subjects (dose confirmation phase) to provide a cohort of 12 subjects at that dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NanoPac® 6 mg/mL (Experimental): NanoPac® 6 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume
  Interventions: Drug: NanoPac®
- NanoPac® 10 mg/mL (Experimental): NanoPac® 10 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume
  Interventions: Drug: NanoPac®
- NanoPac® 15 mg/mL (Experimental): NanoPac® 15 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume
  Interventions: Drug: NanoPac®

INTERVENTIONS:
Drug: NanoPac® — Subjects with prostate cancer scheduled for prostatectomy will have NanoPac® injected intratumorally under image guidance directly into the lobe of the prostate with the dominant lesion 4 weeks prior to prostatectomy.
  Other Names: Paclitaxel

SUMMARY:
Open-label, dose rising, Phase IIa trial of intratumorally-injected NanoPac® 6, 10, or 15 mg/mL in subjects with prostate cancer scheduled for prostatectomy.

DETAILED DESCRIPTION:
In this open-label, dose rising, Phase IIa trial with an expanded cohort at the dose of NanoPac® determined to have the best tolerability and safety profile, subjects with prostate cancer scheduled for prostatectomy will have NanoPac® injected under image guidance directly into the lobe of the prostate with the dominant lesion 4 weeks prior to prostatectomy. The study will include a dose escalation phase and a dose confirmation phase.

In the dose escalation phase, NanoPac® concentrations of 6, 10, and 15 mg/mL in an injection volume of 20% of the lobe of the prostate containing the dominant lesion will be studied in cohorts of 3, with cohorts enrolled sequentially starting at the lowest concentration. Following DSMB review of the cohort data the next cohort may begin enrolling, or an additional 3 at the current dose may be enrolled, or if the first dose does not provide adequate safety and tolerability the study may be halted. The dose determined to be the most suitable for further evaluation, defined as the highest dose with an acceptable safety and tolerability profile as determined by the DSMB, will enroll additional subjects to provide a cohort of 12 subjects at that dose level.

Tumor volume and serum prostate-specific antigen (PSA) will be determined prior to NanoPac® injection. Pharmacokinetic samples, PSA, and ejaculate will be collected in the interval between injection and prostatectomy. Imaging with mpMRI will be performed prior to NanoPac® injection and prior to prostatectomy. Prostate and pelvic lymph nodes excised at prostatectomy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male; 18 years of age and older
* Histopathologically proven adenocarcinoma, Gleason grade ≥ 7 of the prostate planned radical prostatectomy; appropriate for treatment with paclitaxel therapy
* ECOG of 0 or 1
* Laboratory requirements:

  * WBC >2500/mm3
  * Neutrophil >1500/mm3
  * Hemoglobin >10 mg/dL
  * Platelet >100,000/ mm3
  * AST and ALT <2.5 x ULN
  * Total bilirubin <1.5 x ULN
  * Creatinine <2 mg/dL
  * Normal PT/INR and PTT;
* Willing to use appropriate contraception from time of NanoPac® injection until prostatectomy
* Willing to receive an mpMRI

Exclusion Criteria:

* Evidence of locally advanced or metastatic disease;
* Prostate size ≥ 50 cc
* Prior prostatectomy
* Anticipated use of concomitant chemotherapy (other than the protocol specified agents), immunotherapy, or systemic use of hormonal therapy (such as GnRH analogs, antiandrogens, androgen receptor inhibitors, and 5-α reductase inhibitors) prior to surgery
* Treatment with a prior investigational agent within 30 days of first dose of investigational medication
* Any previous local treatment of the prostate (i.e. radiation)
* Any other condition (e.g. psychiatric disorder) that, in the opinion of the Investigator, may interfere with the patient's ability to comply with the study requirements or visit schedule
* Known sensitivity to any of the study medication components
* History of prior malignancy that has not been in remission for >5 years, with the exception of basal cell or squamous cell carcinoma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh Verco, PhD, Study Director — US Biotest, Inc.
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NanoPac® 6 mg/mL: NanoPac® 6 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume 4 weeks prior to prostatectomy.
- NanoPac® 10 mg/mL: NanoPac® 10 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume 4 weeks prior to prostatectomy.
- NanoPac® 15 mg/mL: NanoPac® 15 mg/mL injected into the prostate lobe containing the dominant lesion at a volume of 20% prostate lobe volume 4 weeks prior to prostatectomy.
Period: Overall Study
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Started | 3 | 3 | 10
Completed | 3 | 3 | 9
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL | Total
Number analyzed (Participants) | 3 | 3 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.3) | 73.3 (7.8) | 63.8 (7.9) | 65.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 2 | 1 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 2 | 8 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Treatment Emergent Adverse Events included laboratory assessments, physical examination findings, and vital signs.
Time Frame: Day 1 to Day 29
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
Participants
  All TEAEs | 3 | 2 | 6
  Possibly Related TEAEs | 3 | 0 | 1

2. Secondary Outcome: Tumor Response Based on Change in Image Volume on mpMRI
Description: Tumor response to treatment with NanoPac was determined by evaluating the change in image volume with multiparametric MRI (mpMRI) within three months prior to consent and again within 48 hours of the prostatectomy procedure (Day 29). In those cases where two dimensions/axes were available, width was imputed to height for the purposes of calculation, i.e. the lesion was assumed to be an oblate spheroid. In those cases where only one dimension/axis was available, that dimension/axis was imputed for all three dimensions i.e. the lesion was assumed to be a sphere. For this reason, analyses were performed for all subjects with two dimensions available, as well as those for which at least one dimension was available. The data presented for this outcome measure is the one dimension lesion volume calculation: Lesion Volume (cc) = (3.14/6)*(length)³, where length is the longer or only measured dimension.
Time Frame: Up to three months prior to consent and Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 9
cc
  Lesion Volume at Screening | 3.19 (1.46) | 0.89 (0.44) | 4.89 (5.12)
  Lesion Volume at Day 29 | 1.80 (0.98) | 1.91 (1.50) | 5.10 (7.79)

3. Secondary Outcome: Tumor Response Based on Histologic Evaluation of Biopsied Prostate Samples (Gleason Score)
Description: Prostate tissue samples were obtained via biopsy at baseline and immediately prior to prostatectomy (Day 29). Histologic evaluation of these samples was used to determine the Gleason score, and the results at baseline and Day 29 were used to evaluate the tumor response to treatment with NanoPac®. The Gleason score is calculated by adding together the two grades of cancer cells that make up the largest areas of the biopsied tissue sample. The Gleason score usually ranges from 6 to 10. The lower the Gleason score, the more the cancer cells look like normal cells and are likely to grow and spread slowly; a higher Gleason score is likely to indicate a worse outcome. The Gleason score is used to help plan treatment and determine prognosis.
Time Frame: Screening and Day 29
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
score on a scale
  Gleason Score at Screening | 7.7 (1.2) | 7.0 (0.0) | 7.4 (0.7)
  Gleason Score at Day 29 | 7.7 (1.2) | 7.0 (0.0) | 7.1 (0.9)

4. Secondary Outcome: Percentage of Sample Considered Adenocarcinoma
Description: Tissues excised from the primary tumor during prostatectomy (Day 29) were evaluated for the percentage considered adenocarcinoma
Time Frame: Day 29 (prostatectomy)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of sample adenocarcinoma
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
percentage of sample adenocarcinoma
  Primary Tumor at Screening | 53.3 (5.8) | 33.3 (24.7) | 47.5 (22.0)
  Primary Tumor at Day 29 | 25.0 (15.0) | 56.7 (25.2) | 42.5 (28.0)

5. Secondary Outcome: Concentration of Paclitaxel in the Systemic Circulation
Description: Pharmacokinetic samples were taken on Day 1 at 1, 2, 4, and 6 hours post-injection, and weekly until prostatectomy. All numeric paclitaxel concentration data above the Lower Limit of Quantitation (25 pg/mL) was tabulated by cohort.
Time Frame: Day 1, Day 8, Day 15, Day 22, and Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Plasma paclitaxel concentration (pg/mL)
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
Plasma paclitaxel concentration (pg/mL)
  Day 1 - 1 hr Post-Injection | 5590.00 (2312.336) | 19673.33 (20736.445) | 19010.50 (15105.857)
  Day 1 - 2 hr Post-Injection | 3483.33 (1851.657) | 9103.33 (7881.982) | 12948.70 (10230.061)
  Day 1 - 4 hr Post-Injection | 2240.00 (756.241) | 4740.00 (3889.884) | 6830.80 (5219.617)
  Day 1 - 6 hr Post-Injection | 1926.67 (823.549) | 5006.67 (4938.181) | 5109.00 (3544.025)
  Day 8 | 177.10 (102.777) | 234.33 (73.446) | 404.25 (221.326)
  Day 15 | 65.10 (24.974) | 82.85 (7.283) | 106.11 (62.626)
  Day 22 | 55.70 (15.556) | 43.05 (16.051) | 86.63 (52.358)
  Day 29 | 35.45 (14.496) | 54.75 (36.275) | 57.64 (29.269)

6. Post Hoc Outcome: Change in PSA Density
Description: PSA density was measured with mpMRI
Time Frame: Screening and Day 29
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL/cc
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
ng/mL/cc
  PSA Density at Screening | 3.64 (5.75) | 0.23 (0.02) | 0.31 (0.31)
  PSA Density at Day 29 | 1.95 (2.84) | 0.20 (0.01) | 0.20 (0.11)

7. Post Hoc Outcome: Change in PI-RADS Score
Description: The Prostate Imaging Reporting and Data System (PI-RADS) assessment uses a five-point scale based on the probability that a combination of mpMRI findings on T2 weighting (T2W), Diffusion Weighted Imaging (DWI), and Dynamic Contrast Enhancement (DCE) correlates with the presence of a clinically significant cancer in the prostate gland. A PI-RADS score of 1 is considered to be most probably benign and a score of 5 is considered to be highly suspicious of a prostate malignancy. PI-RADS 1: very low (clinically significant cancer is highly unlikely to be present); PI-RADS 2: low (clinically significant cancer is unlikely to be present); PI-RADS 3: intermediate (presence of clinically significant cancer is equivocal); PI-RADS 4: high (clinically significant cancer is likely to be present); PI-RADS 5: very high (clinically significant cancer is highly likely to be present).
Time Frame: Screening and Day 29
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
Participants
  PI-RADS 3 : Screening | 1 | 1 | 1
  PI-RADS 3 : Day 29 | 0 | 0 | 2
  PI-RADS 4 : Screening | 0 | 1 | 5
  PI-RADS 4 : Day 29 | 1 | 2 | 2
  PI-RADS 5 : Screening | 2 | 1 | 4
  PI-RADS 5 : Day 29 | 2 | 1 | 6

8. Post Hoc Outcome: Tumor Invasion Into Surrounding Tissues
Description: Assessed histologically after TRUS biopsy at Screening and on Day 29 prior to prostatectomy.
Time Frame: Screening and Day 29
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 10
Participants
  Any invasion at Screening? Yes | 2 | 0 | 4
  Any invasion at Screening? No | 1 | 3 | 6
  Any invasion at Day 29? Yes | 2 | 2 | 2
  Any invasion at Day 29? No | 1 | 1 | 8

ADVERSE EVENTS:
Time Frame: 28 days, from Day 1 (the day of NanoPac injection) to Day 29 (the day of prostatectomy)
Description: Adverse events (AEs) were collected at all study visits from the time of dosing. Subjects were required to spontaneously report any AE. Study personnel asked open-ended questions to obtain information about AEs at every visit.
Arm/Group | NanoPac® 6 mg/mL | NanoPac® 10 mg/mL | NanoPac® 15 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoPac® 6 mg/mL (N=3) | NanoPac® 10 mg/mL (N=3) | NanoPac® 15 mg/mL (N=10)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Leucocystosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Procalgia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (5) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Viral URTI (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03077659/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03077659/SAP_001.pdf